CLINICAL TRIAL: NCT02427425
Title: Effectiveness of Transcutaneous Electrical Nerve Stimulation in Patients With Acute Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Vaneska da Graça Cruz Martinelli Lourenzi, Physiotherapist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 1308/09
Record Dates: First submitted 2015-03-10; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Low Back Pain
Keywords: Transcutaneous Electric Nerve Stimulation; Pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TENS group (Experimental): It was applied conventional TENS with FIV effect, frequency of 100 Hertz, a pulse width of 60μs and intensity adjusted according to the individual baseline for each patient without causing muscular contraction. The electrodes were arranged in a cross shape in the paravertebral region (levels T12-L1 and L5 - S1). Treatment consisted of 10 sessions (2x / week / 5 weeks), with each session lasting 30 '.
  Interventions: Device: TENS
- Placebo group (Placebo Comparator): In Placebo group the same procedures of the TENS group were adopted, but did not occur electrical stimulus.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS

SUMMARY:
Introduction: Low back pain is one of the most common complaints in doctors' offices, and acute low back pain is characterized by episodes of pain with less than three weeks duration. The transcutaneous electrical nerve stimulation (TENS), based on the gate control theory of pain proposed by Melzack and Wall in 1965, has been used as an adjunctive therapy in the control of back pain, being a non-invasive, low cost, safe and easy to apply. No studies were found regarding the effectiveness of TENS in acute low back pain.

Objective: To evaluate the effectiveness of TENS in pain management of patients with acute low back pain.

Material and Methods: A randomized clinical trial, double-blinded and placebo-controlled. Patients were selected in the clinics of Federal de University of Sao Paulo (UNIFESP) according to the following criteria: acute low back pain, both genders, aged between 18 and 65 years, pain between 4 and 8cm in pain numeric scale (PNS) and who agreed to participate in the study. After signing the informed consent patients were randomly allocated into one of the groups: TENS group (TG) or Placebo Group (PG). In TG was applied conventional TENS with frequency and intensity variation (FIV) effect, frequency of 100 hertz, a pulse width of 60μs and intensity adjusted according to the individual baseline for each patient without causing muscular contraction. The electrodes were arranged in a cross shape in the paravertebral region (levels T12-L1 and L5 - S1). In PG the same procedures were adopted, but did not occur electrical stimulus. Patients were informed that they could or could not feel electric shocks. Treatment consisted of 10 sessions (2x / week / 5 weeks), with each session lasting 30 '. Assessments were made at the following times: T0 (baseline), T1 to T10 (the beginning and end of each session), T11 (after the last session), T30 (30 days after the last session) and T60 (60 days after the last session). Assessment tools: PNS for pain, short-form 36 (SF-36), Roland-Morris, self-assessment of improvement ("Likert" scale) and drug consumption (daily).

ELIGIBILITY:
Inclusion Criteria:

* acute low back pain
* both genders
* aged between 18 and 65 years
* pain between 4 and 8cm in PNS (pain numeric scale)
* who agreed to participate in the study.

Exclusion Criteria:

* Patients with pain of inflammatory, neoplastic or infectious origin,
* with cardiac pacemaker,
* previous back surgery,
* signs of irritation of nerve roots,
* vertebral fracture, which changed the physical activity in the last three months,
* and pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in pain assessed by visual analog scale | Baseline; 1,2,3,4,5,6,7,8,9,10; 30 and 60 days

SECONDARY OUTCOMES:
Change in functional capacity assessed by the Roland Morris questionnaire | Baseline; 10; 30 and 60 days
Change in self-assessment of improvement assessed by a likert scale | Baseline; 10; 30 and 60 days
Change in Quality of life assessed by the SF-36 questionnaire | Baseline; 10; 30 and 60 days
Change in Drug consumption assessed by the number of NSAIDs consumed | Baseline; 10; 30 and 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Vaneska GC Lourenzi, Principal Investigator — Federal University of São Paulo